CLINICAL TRIAL: NCT07103265
Title: Developing a New Low-intensity Focused Ultrasound (LIFU) Neuromodulation Method to Suppress Tremor
Brief Title: Developing a New LIFU Neuromodulation Method to Suppress Tremor
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REB22-1437
Record Dates: First submitted 2025-07-02; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: We use an in-house developed focused ultrasound system that uses a 128-element phased array transducer (diameter of 135 mm, F#=0.8) operating at 700 kHz and mounted on a specialized arm for stereotactic neuronavigation. Patients will be seated comfortably in a chair equipped with neuronavigation (BrainSight, Rogue) positioning the custom transcranial ultrasound (TUS) array. The TUS array will be applied to the scalp, with ultrasound gel applied, and held in place using the neuronavigation arm. The control session will have the same duration of the real stimulation session, i.e., it will be divided in two 40-minutes long rounds. During the first round, participants will receive sham stimulation which is unfocused, thereby providing the same sound but without sufficient intensity at any location. After the break, during the second round participants will receive TUS stimulation at the same energy parameters as in the real stimulation session but positioning the focus in the CSF space.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real stimulation (Experimental): We use an in-house developed focused ultrasound system that uses a 128-element phased array transducer (diameter of 135 mm, F#=0.8) operating at 700 kHz and mounted on a specialized arm for stereotactic neuronavigation. It has been tested in normal subjects targeting cortical structures (REB#19-1614, #21-0959), and in thalamus for the pilot data collection for this project (REB#22-1437).
  Patients will be seated comfortably in a chair equipped with neuronavigation (BrainSight, Rogue) positioning the custom LIFU array. The LIFU array will be applied to the scalp, with hair parted and ultrasound gel applied, and held in place using the neuronavigation arm.
  Interventions: Device: Transcranial focused ultrasound stimulation
- Sham stimulation (Sham Comparator): Same setting as Real stimulation, but without delivering any ultrasound stimulation.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcranial focused ultrasound stimulation — Parameters Range of values Fundamental frequency 250 kHz Transducer diameter 15 cm Focal distance 13.5 cm (steerable +/- 5-10 mm from the center) Pulse repetition frequency 100 Hz Duty cycle 10% Duration 2 min for each of the 7 foci Peak spatial intensity (Isppa) 10.0 W/cm2 Peak temporal average intensity (Ispta) 1.2 W/cm2 Mechanical index (MI) 0.48 * Thermal index (TI) 0.8oC **
  Arms: Real stimulation
Device: Sham stimulation — Same set-up as for real stimulation but with without delivering any ultrasound stimulation
  Arms: Sham stimulation

SUMMARY:
The investigators aim to apply low intensity focused ultrasound neuromodulation to patients with essential tremor to evaluate the efficacy of this intervention in reducing the amplitude of hand tremor compared to sham stimulation.

DETAILED DESCRIPTION:
Transcranial ultrasound stimulation is a non-invasive brain stimulation that uses low intensity focused ultrasound (LIFU) to modulate neural activity with high spatial precision (Zadeh et al., 2024). Several human and animal studies have demonstrated that LIFU can produce lasting neuromodulatory effects, including both excitatory and inhibitory responses in the primary motor cortex (Zadeh et al., 2024). Furthermore, evidence suggests that LIFU is capable of inducing plasticity in the human brain that resembles long term potentiation or long-term depression (Zeng et al., 2024). The ability of LIFU to induce bidirectional effects, either excitatory or inhibitory, depending on sonication parameters, offers a level of flexibility in tailoring neuromodulatory interventions to individual patient needs and specific neural circuit dysfunctions. Combined with real-time neuronavigation and acoustic modeling tools, LIFU provides a promising platform for precise, personalized, and non-invasive brain stimulation. The modulatory effect of LIFU depends on sonication parameters such as frequency, attenuation, and pulse repetition frequency (Zeng et al., 2024; Manuel et al., 2020), and evidence from both preclinical and clinical studies suggests these effects can persist beyond the stimulation period consistent with long-term potentiation or long-term depression-like plasticity mechanisms (Fomenko et al., 2020; Zadeh et al., 2024).

Unlike other neuromodulatory techniques such as transcranial magnetic stimulation and transcranial direct current stimulation, LIFU offers the unique capability to reach deep brain structures while maintaining a focal spatial resolution. This advantage of precise targeting of deep brain regions such as the thalamus without the need for surgical intervention make LIFU a highly useful modality for investigating disorders (Legon et al., 2018). Structures like the ventral intermediate nucleus (Vim) of the thalamus, commonly implicated in movement disorders such as essential tremor and Parkinson's disease, can be non-invasively stimulated using LIFU to modulate aberrant neural activity.

In a previous study, we piloted an ultrasound transducer integrated with standard optical tracking-based neuro-navigation to establish a safety and tolerability benchmark for LIFU to reduce tremor in patients with Essential Tremor or Parkinson's disease, while also optimizing stimulation parameters prior to broader clinical application. Our open label study, currently under review for publication, demonstrated high efficacy and safety of our system to transiently reduce, in the short term, tremor amplitude measured using accelerometric recordings. By integrating rigorous screening, controlled stimulation parameters, and standardized monitoring protocols, we propose here a randomized sham-controlled study to advance knowledge on efficacy and safety of this technology in a larger clinical sample of patients with these diagnoses. As LIFU continues to expand into therapeutic realms, such foundational research will be essential for supporting its evidence-based integration into neuroscience and medicine.

Objectives. AIM: To determine if we can low intensity focused ultrasound (LIFU, a neuromodulatory form of ultrasound) in the laboratory setting can transiently suppress tremor when targeting motor thalamus in patients with tremor.

HYPOTHESIS: Specific LIFU patterns applied to deep thalamic targets will transiently induce reduce tremor in patients with tremor.

IMPACT: If successful, we could use LIFU to help predict potential efficacy of permanent lesioning on tremor as well as support further investigation of LIFU as a novel non-invasive neuromodulation strategy for tremor.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosis of Essential Tremor OR Diagnosis of Parkinson's Disease

Exclusion Criteria:

* Presence of any neurological diagnosis other than Essential Tremor and Parkinson's Disease
* Family history of Essential Tremor OR Parkinson's Disease
* Inability to undergo MRI or attend to the experimental study sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in power spectral density (PSD) of tremor accelerometric trace between post-sonication (Round 1) and baseline | 5 minutes
  This outcome will be measured using triaxial accelerometry performed on the participants' index finger (treated side). Accelerometry will be analyzed by summing traces from each axis, after using Welch's method to calculate the power spectral density (PSD), with 3-7 Hz tremor frequency range selected for the area under the curve and transformed into logarithmic scale to account for the variability in tremor amplitude at baseline. The primary endpoint will be the percent change in PSD between the post-sonication recording after the 1st Round of the session and the baseline recording.

SECONDARY OUTCOMES:
Change in power spectral density (PSD) of tremor accelerometric trace between post-sonication (Round 2) and baseline | 5 minutes
  This outcome will be measured using triaxial accelerometry performed on the participants' index finger (treated side). Accelerometry will be analyzed by summing traces from each axis, after using Welch's method to calculate the power spectral density (PSD), with 3-7 Hz tremor frequency range selected for the area under the curve and transformed into logarithmic scale to account for the variability in tremor amplitude at baseline. The primary endpoint will be the percent change in PSD between the post-sonication recording after the 2nd Round of the session and the baseline recording.
Change in Clinical Rating Scale for Tremor sub-score corresponding to the sum of scale items related to the treated side between the post-sonication rating and the baseline rating (participants with ET) | 5 minutes
  This applies only to participants with a diagnosis of Essential Tremor
Change in the Movement Disorders Society-Unified Parkinson's Disease Rating Scale sub-score corresponding to the sum of resting tremor items of the scale between the post-sonication rating and the baseline rating (participants with PD). | 5 minutes
  This applies only to participants with a diagnosis of Parkinson's disease